CLINICAL TRIAL: NCT03234335
Title: A Prospective, Non-interventional, Multinational Study Evaluating the Efficacy and the Safety of High Dose Therapy Followed by Autologous Hematopoietic Stem Cell Transplantation as a Frontline Therapy for Myeloma Patients With Severe Renal Impairment (IRMYG Study)
Brief Title: High Dose Therapy Followed by Autologous Transplantation for Myeloma Patients With Severe Renal Impairment
Acronym: IRMYG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0702; 2017-A02180-53 (Other: ANSM)
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Multiple Myeloma; Renal Failure
Keywords: Multiple Myeloma; Renal Failure; Autologous Hematopoietic Stem Cell Transplantation (ASCT); Melphalan
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myeloma patients with severe renal impairment: Myeloma patients with severe renal impairment. Data collection will concern myeloma patients with severe renal impairment who are susceptible to undergo autologous transplantation.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Myeloma patients with severe renal impairment who are susceptible to undergo autologous transplantation will be followed in this study, and data related to the pathology, treatments and transplantation will be reported.

SUMMARY:
Multiple myeloma (MM) is a malignant plasma cell disorder, characterized by the presence of more than 10 % of clonal plasma cells in the bone marrow. Therapeutic intervention is recommended when at least one of the myeloma defining events occurs (CRAB features). Renal impairment (RI) is one of the most common complications of MM, accounting for 20-30 % of MM patients at diagnosis and 40-50% of patients during the course of their disease. To date, there is no defined consensus for the management of myeloma patients with renal failure. It is then of clinical importance to better considering available therapeutic options to improve responses and survival of these patients.

DETAILED DESCRIPTION:
RI is associated with poor prognosis and short median survival (32 months vs 55 months for MM patients with normal renal function). Thus, RI remains a major challenge for hematologists, including decisions on optimal anti-myeloma therapy, potential dialysis, supportive care and quality of life. The combination of a proteasome inhibitor and an immunomodulator is the preferred induction treatment for newly diagnosed transplant-eligible MM patients. After induction, high-dose therapy with Autologous Stem Cell Transplant (ASCT) is the standard of care for these patients. However, concerns related to management of comorbidities and treatment side effects question about therapeutic options for patients with severe renal damage. Of interest, recent studies argued that high-dose therapy followed by ASCT could be a feasible and safe method for renal failure MM patients. Yet, these observations on small sample size patients groups need to be confirmed with standardized conditions. This study proposes to evaluate the efficacy and the safety of this therapeutic strategy in MM patients with severe renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 66 years-old
* Patients with symptomatic, measurable and newly diagnosed multiple myeloma associated:
* Severe renal failure at the time of transplantation (creatinine clearance < 40 ml/min/1.73m², CKD-EPI: Chronic Kidney Disease Epidemiology Collaboration)
* Partial response after induction treatment
* For patients who undergo autologous transplantation, absence of known contraindication for transplantation
* Absence of amylose
* Patient affiliated to a social security regimen or beneficiary of the same
* Signed written informed consent form

Exclusion Criteria:

* Patient without at least a partial hematological response following the induction stage
* Medical history of previous malignancy
* Patient under guardianship or deprived of his liberty or any condition that may affect the patient's ability to understand and sign the informed consent (art. L.1121-6, L.112-7, L.1211-8, L.1211-9)
* Pregnant or breastfeeding woman
* Declining participation

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Myeloma patients with severe renal impairment suseptible of undergoing autologous transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Non Relapse Mortality post-transplantation | 100 days post-transplantation
  Non-relapse mortality at Day +100 post-transplantation will be reported.

SECONDARY OUTCOMES:
Overall survival | 2 years post-transplantation
  Overall survival at 2 years post-transplantation will be reported.
progression-free survival | 2 years post-transplantation
  progression-free survival at 2 years post-transplantation will be reported.
Number of toxicities | 2 years post-transplantation
  Number of hematological and extra-hematological toxicities linked to autologous stem cell transplantation will be reported during 2 years.
presence of hematological response | 6 months
  The presence of hematological response at Day+100 and at 6 months post-transplantation will be reported.
Level of renal response | 3 months, 6 months and one year
  Level of renal response at 3 months, 6 months and one year post-transplantation will be quantified and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Cornillon, MD, Principal Investigator — CHU de Saint-Etienne
Locations (33):
- Algeria (2):
  - Centre Pierre et Marie Curie, Algiers
  - EHU Oran, Oran
- CHU Sart Tilman, Liège, Belgium
- France (29):
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier d'Argenteuil, Argenteuil
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre Hospitalier de Boulogne, Boulogne
  - CHU de Brest, Brest
  - Centre Hospitalier Universitaire de Caen, Caen
  - Centre Hospitalier de Cholet, Cholet
  - Centre Hospitalier Universitaire de Clermont Ferrand, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Hôpital Saint-Eloi, Montpellier
  - Centre Hospitalier Universitaire de Nancy, Nancy
  - Hôpital Archet, Nice
  - Institut Curie, Paris
  - Groupe Hospitalier Pitié-Salpétrière, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Tenon, Paris
  - Hôpital Cochin, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Saint-Bernard, Poitiers
  - CHU de Rennes, Rennes
  - Hôpital Victor Provo (Roubaix), Roubaix
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - Centre Hospitalier de Saint Quentin, Saint-Quentin
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
- American University of Beirut, Beirut, Lebanon